CLINICAL TRIAL: NCT06210243
Title: A Single-arm, Open-label Clinical Study to Assess the Safety and Efficacy of the C752 CAR-T Cells for Patients With CD19+ Refractory/Relapsed B Cell Non-Hodgkin Lymphoma
Brief Title: C752 for Refractory/Relapsed B Cell Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the PI's determination
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Collaborators: Shanghai PerHum Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH02001
Record Dates: First submitted 2024-01-07; First posted 2024-01-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Lymphoma, B-Cell; CAR-T
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C752 (Experimental)
  Interventions: Biological: C752

INTERVENTIONS:
Biological: C752 — C752 will be administered on Day 0

SUMMARY:
It is a single-arm, open-label clinical study to assess the safety and efficacy of the C752 CAR-T Cells for patients with CD19+ refractory/relapsed B cell non-Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with federal, local, and institutional guidelines, Males and females ≥18 years of age at the time of consent
* Documented diagnosis of Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
* Have progression by least one systemic treatment and no available standard of care treatment.
* At least one measurable lesion by Lugano 2014
* Expected survival ≥ 12 weeks
* Have an ECOG performance status of 0 or 1
* Adequate organ function
* Screening test indicates histopathological CD19 + if the subject received CD19-targeted therapy
* Women of childbearing age must have a negative pregnancy test, and agree to take effective contraception during the trial

Exclusion Criteria:

* Treatment with any prior HSCT, gene therapy product, cell therapy product ect.
* Central nervous system involvement
* HBV/HCV
* HIV infection
* Concurrent use of systemic steroids or immunosuppression
* Uncontrolled active infection
* Wash-out period of from the last anti-cancer treatment
* Active second malignancy
* Have not recovered from the effects of previous therapy
* Have psychological or physical conditions that do not permit compliance with the protocol
* Pregnant or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-12-24 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of adverse events (AEs) | 1 year
Dose Limiting Toxicities | First 28 days s after C752 injection

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1 year
  Objective response rate after C752 injection as defined by Lugano 2014
PFS | 1 year
Pharmacokinetic - AUC | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, M.D., Principal Investigator — 920th Hospital
Locations (1):
- 920th Hospital of Joint LogisticsSupport Force of People's Liberation, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No